CLINICAL TRIAL: NCT02096341
Title: A Phase 1 Pilot Study of the Subcutaneous (s.c.) Route to Facilitate the Administration of RRx-001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Subcutaneous administration of RRx-001 is no longer of interest.
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-12-01
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Malignant Solid Tumor; Lymphomas
MeSH Terms: conditions — Lymphoma | interventions — RRx-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RRx-001 (Experimental): RRx-001 will be administered as subcutaneous injections twice weekly for at least 8 weeks. At least three subjects must complete 2 weeks of treatment with RRx-001 at each dose level, before escalation to the next higher RRx-001 dose level; 2 doses-16 and 27 mg/m2- will be tested.
  Interventions: Drug: RRx-001

INTERVENTIONS:
Drug: RRx-001 — RRx-001 Dose level 1 (16 mg/m2) twice weekly
  RRx-001 Dose level 2 (27 mg/m2) twice weekly

SUMMARY:
To investigate the dosage of RRx-001 by the subcutaneous route.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-escalation study of RRx-001. Subjects will receive RRx-001 administered as subcutaneous injections twice weekly for at least 8 weeks. At least three subjects must complete 2 weeks of treatment with RRx-001 at each dose level, before escalation to the next higher RRx-001 dose level; 2 doses-16 and 27 mg/m2- will be tested.

The purpose of the study is to extend the dosage options for RRx-001 since faster subcutaneous (SC) administration may increase convenience versus the traditional IV method. The study also will also measure the mean concentrations of an RRx-001 metabolite in the blood (pharmacokinetics; PK) versus the IV formulation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* ECOG (performance) status of 0, 1 or 2.
* Histologically or cytologically confirmed primary or metastatic advanced solid tumors or lymphoma. Subjects with curative treatment options are not eligible for the protocol.
* No active ongoing cancer treatment (except for prostate cancer subjects receiving luteinizing hormone-releasing hormone (LHRH) agonists and anti-androgens such as; Flutamide, Dutasteride, and Finasteride).
* Adequate organ and bone marrow function.
* Male and female subjects of childbearing potential must agree to use contraception.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Use of anti-coagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 10 weeks

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of RRx-001-glutathione conjugate | 1 day
Peak Plasma Concentration (Cmax) of RRx-001-glutathione conjugate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Infante, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States

REFERENCES:
- See also: EpicentRx, Inc Home page. — http://www.epicentrx.com/